CLINICAL TRIAL: NCT02339779
Title: the Breast Reconstruction With External Pre-expansion and Autologous Fat Transfer Versus Standard Therapy Trial
Brief Title: Breast Reconstruction With External Pre-expansion and Autologous Fat Transfer Versus Standard Therapy
Acronym: BREAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC142059
Record Dates: First submitted 2015-01-07; First posted 2015-01-15 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: fat grafting; fat injection; lipoaspirate; fat transfer; lipofilling; liposculpturing; lipoinjection; lipotransfer; breast reconstruction; external pre-expansion; BRAVA; EVE
MeSH Terms: conditions — Breast Neoplasms | interventions — Breast Implants; Breast Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous fat transfer reconstruction (Experimental): Breast reconstruction achieved by serial autologous fat transfer (AFT) procedures, accompanied by external tissue expansion of the breast.
  Interventions: Procedure: autologous fat transfer
- Reconstruction with breast implants (Active Comparator): Control group will receive implant-based reconstruction, in some cases preceded by the implantation of a tissue expander.
  Interventions: Procedure: breast implant

INTERVENTIONS:
Procedure: autologous fat transfer — Each procedure consists of the transfer of syringe-aspirated fat (form the abdomen, thighs, flanks) to the breast by injection in the subcutaneous planes.
  Typically three separate procedures are needed for a complete breast reconstruction:
  1. First session comprises of sub- and intrapectoral fat transfer during the primary mastectomy surgery, providing volume to the deep tissue planes.
  2. Second session is preceeded by wearing an external pre-expansion device to prepare the recipient site for grafting. It aims to give the breast its shape and initial volume.
  3. Third session is also preceded by external pre-expansion and aims to provide extra volume of the breast to achieve symmetry with the healthy breast.
  Other Names: lipofilling; fat grafting; lipografting; lipoaspirate grafting; autologous fat injection
  Arms: Autologous fat transfer reconstruction
Procedure: breast implant — Implant-based reconstruction typically will occur as follows:
  1. During the primary mastectomy surgery, a tissue expander will be implanted subpectorally.
  2. The tissue expander will be gradually filled with sterile saline during outpatient clinic visits.
  3. When the desired volume is achieved, a second operation will be planned, to exchange the tissue expanded with the definite breast implant.
  (Note: in patients who are receiving encapsulectomy and implant exchange, the first 2 steps are skipped.)
  Other Names: breast prosthesis
  Arms: Reconstruction with breast implants

SUMMARY:
This multicentre randomized controlled trial aims to evaluate a new breast reconstruction technique- autologous fat transfer (AFT). Female patients with breast cancer schedule to receive a mastectomy (or having undergone mastectomy in the past) will be randomized to undergo breast reconstruction with either AFT (intervention group) or reconstruction with implants (control group). AFT will be evaluated in terms of quality of life, aesthetic result, complications, oncological safety and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age of 18 years and older
* History or in candidate for a mastectomy procedure in the near future
* Patients' choice to undergo a breast reconstruction
* Wanting to participate in this study
* Patient is able to wear the BRAVA device

Exclusion Criteria:

* Active smoker or a history of smoking 4 weeks prior to surgery
* Current substance abuse
* History of lidocaine allergy
* History of silicone allergy
* 4 weeks or less after chemotherapy
* History of radiation therapy in the breast region
* Oncological treatment includes radiotherapy after mastectomy
* Kidney disease
* Steroid dependent asthma (daily or weekly) or other diseases
* Immune-suppressed or compromised disease
* Uncontrolled diabetes
* BMI>30
* Large breast size (i.e. larger than cup C), unless the patient prefers reduction of the contralateral side towards Cup C
* Extra-capsular silicone leaking from the encapsulated implant from a previous breast reconstruction
* The treating plastic surgeon has strong doubts on the patient's treatment compliance
* Claustrophobia for an MRI-scan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Breast-related Quality of life (BREAST_Q) | 1 year
  Measured by the BREAST-Q questionnaire (quality of life subdivision) preoperatively and 1 year postoperatively

SECONDARY OUTCOMES:
Aesthetic result | 1 year
  The overall aesthetic result will be measured using 3D-photographs which will be assessed by a panel of independent plastisch surgeons, ex-breast cancer patients and healthy volunteers. In addition, the volume, shape and symmetry will be assessed by the patient using the BREAST-Q questionnaire (satisfaction with breasts subdivisions) at 1 year postoperatively.
Complications | 1 year
  Measurement of short-term als well as mid-term complications associated with procedures as well as (serious) adverse events.
Oncological safety | 5 years
  Oncological follow-up will comply to the guidelines for breast cancer and will take place by a yearly consult with the oncological surgeon (including physical examination and mammography/ultrasound/MRI) for 5 years postoperatively. All (loco)regional and distant recurrences will be recorded and compared between both grops.
Cost-effectiveness | 1 year
  Cost-effectiveness analysis to determine the intramural and socio-economic costs associated with the breast reconstruction treatment. It will be calculated according to the guidelines of the "Instuction manual cost-effectiveness analysis" (Handleiding kostenonderzoek) of the Dutch Health Institute (Zorginstituut Nederland).
Sensibility | 1 year
  Measurement of skin sensitivity with Semmes Weinstein Monofilaments, 12 months after final reconstruction surgery.
Donor site satisfaction | 2 years
  Measurement of quality of life and satisfaction at AFT donor sites, as measured by the BODY-Q questionnaire and additional questions concerning liposuction sites.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Piatkowski de Grzymala, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (7):
- Netherlands (7):
  - Amstelland Hospital, Amstelveen
  - VU Medical Center, Amsterdam
  - Alexander Monro Breast cancer hospital, Bilthoven
  - Amphia Hospital, Breda
  - Ziekenhuis Groep Twente Hospital, Hengelo
  - Maastricht University Medical Centre (MUMC+), Maastricht
  - Bronovo-MCH Hospital, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wederfoort JLM, Trommelen DAX, Al Tarah M, Hommes JE, van Kuijk SMJ, van der Hulst RRWJ, Piatkowski AA; BREAST- trial investigators. Volumetric evaluation of autologous fat transfer for total breast reconstruction. J Plast Reconstr Aesthet Surg. 2024 Dec;99:317-328. doi: 10.1016/j.bjps.2024.09.083. Epub 2024 Sep 29. PMID 39413587
- [Derived] Wederfoort JLM, Schop S, van der Broeck LCA, Hommes JE, van Kuijk SMJ, Timmermans F, Smit JM, Heuts EM, de Wit T, van der Hulst RRWJ, Piatkowski AA. Superior Sensibility after Full Breast Reconstruction with Autologous Fat Transfer. Plast Reconstr Surg. 2024 Feb 1;153(2):316-323. doi: 10.1097/PRS.0000000000010619. Epub 2023 Apr 28. PMID 37114918
- [Derived] Piatkowski AA, Wederfoort JLM, Hommes JE, Schop SSJ, Krastev TK, van Kuijk SMJ, van der Hulst RRWJ; Breast Reconstruction With External Preexpansion & Autologous Fat Transfer vs Standard Therapy (BREAST) Trial Investigators. Effect of Total Breast Reconstruction With Autologous Fat Transfer Using an Expansion Device vs Implants on Quality of Life Among Patients With Breast Cancer: A Randomized Clinical Trial. JAMA Surg. 2023 May 1;158(5):456-464. doi: 10.1001/jamasurg.2022.7625. PMID 36857058
- [Derived] Schop SSJ, Hommes JE, Krastev TK, Derks D, Larsen M, Rakhorst H, Schmidbauer U, Smit JM, Tan T, Wehrens K, de Wit T, van der Hulst RRWJ, Piatkowski de Grzymala AA. BREAST trial study protocol: evaluation of a non-invasive technique for breast reconstruction in a multicentre, randomised controlled trial. BMJ Open. 2021 Sep 16;11(9):e051413. doi: 10.1136/bmjopen-2021-051413. PMID 34531218